CLINICAL TRIAL: NCT03702179
Title: Phase II Trial of Durvalumab (Medi4736) Plus Tremelimumab With Concurrent Radiotherapy in Patients With Localized Muscle Invasive Bladder Cancer Treated With a Selective Bladder Preservation Approach
Brief Title: Durvalumab Plus Tremelimumab With Concurrent Radiotherapy for Localized Muscle Invasive Bladder Cancer Treated With a Selective Bladder Preservation Approach
Acronym: IMMUNOPRESERVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: AstraZeneca (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2017-A-IEC(VEJ)-1
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2023-08

CONDITIONS: Invasive Bladder Cancer
Keywords: localized muscle invasive bladder cancer; bladder preservation; durvalumab; tremelimumab; radiotherapy
MeSH Terms: interventions — durvalumab; tremelimumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: The study will be conducted using a two-stage sequential design. Using the assumption that the treatment would be considered ineffective if it had a response proportion similar to radiotherapy alone (P0: 0.5) but would be of considerable interest if it had a response proportion of 70% of more (P1: 0.7), the sample size requirement is 12 patients for the first stage and 20 additional patients for the second stage. Six or more responses in the first stage were required for continuation to second stage accrual. The study was planned to have a type I error of 0.10 and a power of 80% in a one sided test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab (Experimental): The treatment consisted of initial TUR of the tumor, with multiple random biopsies of normal-appearing bladder urothelium, followed by durvalumab 1500 mg i.v. plus tremelimumab 75 mg i.v., every 4 weeks for a total of 3 doses.
  Two weeks after the initiation of immunotherapy, normofractionated external-beam radiotherapy with high-energy photons will be started. Radiotherapy will be administered concurrently with immunotherapy at doses of 46 Gy to the minor pelvis and 64-66 Gy to the bladder.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab — All patients will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) for up to 3 doses/cycles each, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30kg or below the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W and 1mg/kg tremelimumab Q4W until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500mg plus tremelimumab 75 mg Q4W.
  Other Names: MEDI4736
Drug: Tremelimumab — All patients will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) for up to 3 doses/cycles each, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30kg or below the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W and 1mg/kg tremelimumab Q4W until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500mg plus tremelimumab 75 mg Q4W.
Radiation: Radiotherapy — Radiotherapy at doses of 46 Gy to the minor pelvis and 64-66 Gy to the bladder.

SUMMARY:
Combined-modality treatment of localized muscle invasive bladder cancer including transurethral resection (TUR), radiotherapy and dual checkpoint inhibition immunotherapy could achieve pathological complete response in some patients. These patients could avoid to undergone radical surgery with radical cystectomy and preserve their bladder, without the side-effects associated with chemotherapy and surgery. This study has been design to determine the efficacy of durvalumab plus tremelimumab with concurrent radiotherapy in terms of pathological response rate in patients with localized muscle invasive bladder cancer treated with bladder preservation intent.

DETAILED DESCRIPTION:
The treatment consisted of initial TUR of the tumor, with multiple random biopsies of normal-appearing bladder urothelium, followed by durvalumab 1500 mg i.v. plus tremelimumab 75 mg i.v., every 4 weeks for a total of 3 doses.

Two weeks after the initiation of immunotherapy, normofractionated external-beam radiotherapy with high-energy photons will be started. Radiotherapy will be administered concurrently with immunotherapy at doses of 46 Gy to the minor pelvis and 64-66 Gy to the bladder.

Six weeks after the end of radiotherapy, ALL patients will undergo a new cystoscopy with biopsies of the tumor bed and all residual present lesions as an efficacy determination. In patients with persistent prominent inflammatory reaction at this moment, the cystoscopy can be performed 1-2 weeks later (6 to 8 weeks after the end of radiotherapy). Response is defined as an absence of invasive cancer at post immunotherapy biopsy (≤cT1). Patients with response to immunotherapy will be candidates to bladder preservation, whereas in those with residual muscle invasive tumor the possibility of salvage radical cystectomy must be evaluated. Patients developing an isolated bladder invasive relapse during follow-up will be also possible candidates to salvage cystectomy, whereas those developing a superficial relapse in the preserved bladder will be managed with TUR and intravesical BCG.

Patients will be followed up every 3 months the first year, every 4 months the second year and every 6 months thereafter with abdomen and pelvis CT scan, Rx thorax, urine cytology. Additionally, the mandatory efficacy cystoscopy and bladder biopsy (6w post RT), other cystoscopy and bladder biopsy will be performed in case of detection abnormalities in the cytology or imaging studies. The study will be closed 2 years after the last patient inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed the informed consent prior to undergoing any study procedure.
* Patients must be 18 years of age or older.
* Patients must have Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* A paraffin-embedded tumor sample must be available for the associate molecular study.
* Body weight >30 Kg.
* Adequate normal organ and marrow function.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre- menopausal patients.
* Patient is willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both Sponsor staff and/or staff at the study site).
* Participation in another clinical study with an investigational product during the last 30 days.
* Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Previous treatment with radiotherapy to the bladder, systemic chemotherapy or immune checkpoint inhibitors. Prior intravesical Bacillus Calmette-Guérin (BCG) treatment for non-muscle invasive bladder cancer is allowed, 28 days prior to study.
* Presence of regional lymph node or metastatic extension of the disease.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) <<for durvalumab monotherapy and durvalumab + tremelimumab combination studies this criterion can be removed. For durvalumab ±tremelimumab in combination with an agent with pro-arrhythmic potential or where effect of the combination on QT is not known if this criterion should be retained. Patient safety and the cardiac ECG should be consulted as needed>>.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.

* Any concurrent chemotherapy, investigational product (IP) other than studied in this protocol, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders.
* Uncontrolled intercurrent illness.
* History of another primary malignancy.
* History of active primary immunodeficiency.
* Active infection.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of the investigational medical products (IMP).
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* Known allergy or hypersensitivity to IP or any excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier García del Muro, M.D., Study Chair — Instituto Catalán de Oncología L'Hospitalet
Locations (7):
- Spain (7):
  - Instituto Catalán de Oncología Badalona, Badalona, Barcelona
  - Centro Oncológico de Galicia, A Coruña
  - Instituto Catalán de Oncología L'Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - H.U. Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab + Tremelimumab: The treatment consisted of initial TUR of the tumor, with multiple random biopsies of normal-appearing bladder urothelium, followed by durvalumab 1500 mg i.v. plus tremelimumab 75 mg i.v., every 4 weeks for a total of 3 doses.
  Durvalumab: All patients will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) for up to 3 doses/cycles each, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30kg or below the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W and 1mg/kg tremelimumab Q4W until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500mg plus tremelimumab 75 mg Q4W.
  Tremelimumab: All patients will receive durvalumab (MEDI4736) (1500mg Q4W) in combination with tremelimumab (75 mg IV Q4W) for up to 3 doses/cycles each, unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. If a patient's weight falls to 30kg or below the patient should receive weight-based dosing equivalent to 20 mg/kg of durvalumab Q4W and 1mg/kg tremelimumab Q4W until the weight improves to >30 kg, at which point the patient should start receiving the fixed dosing of durvalumab 1500mg plus tremelimumab 75 mg Q4W.
  Radiotherapy 46 Gy to the minor pelvis and 64-66 Gy to the bladder.
Period: Overall Study
Arm/Group | Durvalumab + Tremelimumab
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 71 [49 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) [Count of Participants; unit: Participants] — Describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working...).
  The scale ranges from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (Dead).
  Participants
    ECOG 0 | 25
    ECOG 1 | 7
Histology [Count of Participants; unit: Participants] — Describes the histology subtype of tumor, the type of cells from which the tumor has arisen.
  Participants
    Urothelial carcinoma | 31
    Mixed urothelial carcinoma | 1
Clinical T stage [Count of Participants; unit: Participants] — T stage according to AJCC criteria. Describes the extent of tumor spread and size. T ranges from T1 (The tumor has spread to the connective tissue but it does not involve the bladder wall muscle) to T4 (The tumor has spread to any of the following: the abdominal wall, the pelvic wall, the prostate or seminal vesicle, or the uterus or vagina).
  Participants
    T2 | 28
    T3 | 3
    T4 | 1
Previous bladder cancer non-muscle invasive [Count of Participants; unit: Participants] — Describes the history of bladder cancer for patients, the presence or not of previous local bladder cancer that may have occured earlier before inclusion and that may be treated with resection of local treatments.
  Participants
    Yes | 14
    No | 18
Previous treatment [Count of Participants; unit: Participants] — Type of previous treatments for bladder cancer before patient inclusion
  Participants
    Bacillus Calmette-Guérin (BCG) | 9
    Mitomycin | 1
    Transurethral Resection of Bladder Tumor (TURBT) | 1
    No treatment | 21
PD-L1 expression [Count of Participants; unit: Participants] — Programmed death-1 ligand 1 (PD-L1) expression levels in tumor tissue samples has been described as correlated with response to immunotherapy such as the experimental treatment studied in this trial. PD-L1 expression is measured by immunohistochemistry in tumor sample and could be positive (high expression) or negative (low expression).
  Participants
    Positive | 15
    Negative | 12
    Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Pathological Response
Description: Pathological response is defined as the absence of muscle- invasive bladder cancer at post-treatment biopsy (≤cT1). Cystoscopy and bladder biopsy six weeks since the end of radiotherapy.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab + Tremelimumab: Experimental arm:
  Durvalumab 1500 mg i.v. plus tremelimumab 75 mg i.v., every 4 weeks for a total of 3 doses Radiotherapy 46 Gy to the minor pelvis and 64-66 Gy to the bladder.
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 28
Participants
  Complete Response (≤T1) | 26
  Non-response (MIBC) | 2

2. Secondary Outcome: Rate of Patients With Bladder Preserved
Description: Number of patients whom bladder has been preserved after cytoscopic evaluation.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 28
Participants
  Preserved bladder | 28
  Not preserved bladder | 0

3. Secondary Outcome: Rate of Immediate Salvage Cystectomies
Description: Number of patients with indication of salvage cystectomies after first trial-related cystoscopic evaluation.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
Participants
  Radical cystectomy performed | 1
  Radical cystectomy not required | 31

4. Secondary Outcome: Rate of Late Salvage Cystectomies
Description: Number of patients with indication of salvage cystectomies based on follow-up cystoscopic evaluation.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
Participants
  Required late cystectomy | 2
  Not required late cystectomy | 30

5. Secondary Outcome: Survival With Bladder Preserved Free of Tumor
Description: Time from the start of immunotherapy to either the date of cystectomy or the date of recurrence of muscle- invasive bladder carcinoma or metastasis.
  Here we report the estimated rate of patients free of event at 24 months after the start of immunotherapy. Estimation by kaplan meier method.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients (%) free of event
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
percentage of patients (%) free of event | 65 [50.3 to 84.1]

6. Secondary Outcome: Disease-free Survival
Description: Time from treatment start to tumour relapse or distant progression (without Salvage cystectomy). Bladder relapse with salvage cystectomy is not considered as an event.
  Deaths are also considered as events. Here we report the estimated rate of patients free of events at 24 months after the start of the immunotherapy. Estimation by kaplan meier method.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients (%) free of event
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
percentage of patients (%) free of event | 71.4 [57.2 to 89.1]

7. Secondary Outcome: Overall Survival
Description: Time from the start of immunotherapy to the date of death due to any cause. The reported outcome is the estimated ratio of patients alive at 24 months after start of immunotherapy using kaplan meier method.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients (%) alive
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
percentage of patients (%) alive | 84.3 [72.5 to 97.9]

8. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Frequency, nature and number of patients developing adverse events throughout follow up
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 32
Participants
  Treatment related adverse events of any grade: Had treatment-related adverse events | 31
  Treatment related adverse events of any grade: Had not treatment-related adverse events | 1
  Treatment related adverse events Grade ≥3: Had treatment-related adverse events | 10
  Treatment related adverse events Grade ≥3: Had not treatment-related adverse events | 22

ADVERSE EVENTS:
Time Frame: Throughout the study period, approximately a median o 24 months follow up.
Arm/Group | Durvalumab + Tremelimumab
All-Cause Mortality (participants affected / at risk) | 7/32
Serious Adverse Events (participants affected / at risk) | 11/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab + Tremelimumab (N=32)
Fever (General disorders) | 3
Immunomediated colitis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify - (Respiratory, thoracic and mediastinal disorders) | 2
Acute pyelonephritis (Renal and urinary disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Hypotension (Vascular disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Fecaloid peritonitis (Gastrointestinal disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab + Tremelimumab (N=32)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 15
Diarrhea (Gastrointestinal disorders) | 9
Urinary frequency (Renal and urinary disorders) | 11
Hyperthyroidism (Metabolism and nutrition disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 5
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Urinary tract pain (Renal and urinary disorders) | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Hypothyroidism (Metabolism and nutrition disorders) | 4
Hematuria (Blood and lymphatic system disorders) | 4
General disorders and administration site conditions - Other, specify (General disorders) | 3
Aspartate aminotransferase increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Insomnia (General disorders) | 3
Edema limbs (General disorders) | 3
Dizziness (Nervous system disorders) | 3
Constipation (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03702179/Prot_SAP_000.pdf